CLINICAL TRIAL: NCT05353309
Title: Iliac Angioplasties: Impact of the Fusion of Images on the Irradiation Rate
Acronym: AIFITI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: European Clinical Trial Experts Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-A03414-35
Record Dates: First submitted 2022-04-05; First posted 2022-04-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Irradiation Rate; Image, Body; Iliac Artery Disease
Keywords: irradiation patient rate; iliac angioplasty
MeSH Terms: interventions — Angioplasty

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Angioplasty DSA (Active Comparator): Reference procedure (DSA), comprising: production of fluoroscopy images for placement of endoluminal material and navigation, subtracted angiography with placement of flaps to reduce the field of rays ("collimation ") for visualization of the arterial axis (in low dose, pulsed with maximum collimation), the realization of possible oblique incidences (external iliac), the catheterization with or without placement of a post-inflation stent, then the realization of a second subtracted control angiogram.
  Interventions: Procedure: Standard Angioplasty
- Angioplasty DSA+Fusion (Experimental): Procedure under study (DSA+Fusion), including: production of fluoroscopy images for placement of the endoluminal material and navigation, 2 fluoroscopy images specifically for image fusion registration (from the images scanner), selective angiography under fluoroscopy with collimation to improve registration (in low dose mode, pulsed with maximum collimation), if possible no oblique views (3D markers of the fusion), with or without placement of post-inflation stent followed by subtracted control angiography
  Interventions: Procedure: Angioplasty with D images

INTERVENTIONS:
Procedure: Standard Angioplasty — Angioplasty Iliac done following standard practice
  Arms: Angioplasty DSA
Procedure: Angioplasty with D images — Angioplasty Iliac under additional 3D Images merged as surgery support
  Arms: Angioplasty DSA+Fusion

SUMMARY:
Atherosclerosis can cause the arteries to narrow (stenosis) or clog (occlude), leading to reduced blood flow.

Arteriography or angiography is a radiological examination of the arteries which will make it possible to confirm and quantify the severity of the damage to the artery and which, in certain cases, can be directly treated by angioplasty with or without stenting (selective angioplasty).

Digital subtraction angiography (DSA), the reference technique, provides good image quality. The fluoroscopy used today during angioplasty procedures makes it possible to obtain images in real time and to guide the progression of the endovascular material in the arterial axis. Image fusion is an established technique for the endovascular treatment of aortic aneurysms. The feasibility of image fusion for the iliac arterial axes has already been assessed and is reproducible. However, there is no assessment of the irradiation rate in iliac angioplasty, using intraoperative image fusion, compared to standard angioplasty practices.

DETAILED DESCRIPTION:
Atherosclerosis can cause the arteries to narrow (stenosis) or clog (occlude), leading to reduced blood flow. Iliac stenosis can be asymptomatic or symptomatic. Clinical manifestations are related to the degree of narrowing. The symptoms are in order of increasing severity: pain in the legs when walking (intermittent claudication), at rest, even foot or leg ulcers.

Arteriography or angiography is a radiological examination of the arteries requiring the injection of contrast product which will make it possible to confirm and quantify the severity of the damage to the artery and which, in certain cases, can be directly treated by angioplasty with or without stenting (selective angioplasty).

Digital subtraction angiography (DSA), the reference technique, provides good image quality. The fluoroscopy used today during angioplasty procedures makes it possible to obtain images in real time and to guide the progression of the endovascular material in the arterial axis. Image fusion is an established technique for the endovascular treatment of aortic aneurysms. The feasibility of image fusion for the iliac arterial axes has already been assessed and is reproducible. However, there is no assessment of the irradiation rate in iliac angioplasty, using intraoperative image fusion, compared to standard angioplasty practices.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, over the age of 18
* Patient with a primary and/or external iliac lesion (TASC A, B and C)
* Patient for whom unilateral angioplasty is indicated
* Affiliated patient or beneficiary of a social security scheme
* Patient having been informed and having signed a written consent.

Exclusion Criteria:

* Patient with a BMI strictly less than 18.5 or greater than or equal to 30.0 kg/m²
* Patient with long iliac thrombosis (including the primitive iliac and the external iliac)
* Patient with a known allergy to iodine
* Patient with a contraindication related to the procedure
* Patient for whom a bilateral iliac procedure is indicated
* Patient requiring an associated infra-inguinal endovascular procedure
* Patient participating in another clinical study
* Protected patient: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision
* Pregnant, breastfeeding or parturient women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2021-05-25 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Irradiation rate | "immedialtely at the end of surgery procedure"
  mean irradiation rate during iliac angioplasty will be compared between the 2 study groups The primary endpoint of the research is the patient's intraoperative irradiation rate defined by measuring the dose area product (DAP) in Gy.cm2

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU de Nantes, Nantes, Brittany Region
  - Saint Martin Private Hospital, Caen, Normandy

IPD SHARING:
Plan to Share IPD: Undecided